CLINICAL TRIAL: NCT00421070
Title: The Evaluation of Relaxation Massage Therapy as an Intervention Treatment for Reducing the Level of Arousal and Aggression on a Young Adult Psychiatric Inpatient Unit
Brief Title: Effect of Massage Therapy on Aggression in a Psychiatric Inpatient Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Melbourne Health (Other)
Collaborators: National Health and Medical Research Council, Australia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HREC2005.060
Record Dates: First submitted 2007-01-10; First posted 2007-01-11 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Psychiatric &or Mood Disorder
Keywords: Aggression; Massage; Stress; Psychiatric inpatient
MeSH Terms: conditions — Mood Disorders; Aggression | interventions — Massage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment as usual (No Intervention): Observational component
- Intervention (Active Comparator): Massage therapy adjunct comparator
  Interventions: Procedure: Massage therapy

INTERVENTIONS:
Procedure: Massage therapy — A qualified massage therapist will administer a 20-minute standard massage procedure with the client sitting fully clothed in a special massage chair. The massage therapy session will consist of ; 1) long, broad stroking with light-moderate pressure to the back, compression to the back (parallel to spine) from the shoulders to base of spine, trapezius squeeze, finger pressure on the shoulder; 2) arms dropped to the side with arms kneaded from shoulder to lower arm and pressing down on upper and lower arms; 3) entire hands massaged and pulling of fingers, light kneading to area of cervical vertebrae, pressing down on trapezius with finger pressure and squeezing continuing down the arms.
  Arms: Intervention

SUMMARY:
The purpose of this study is to investigate whether relaxation massage therapy is effective in reducing the levels of arousal and aggression on a young adult inpatient unit. It is hypothesised that relaxation massage therapy will lead to a lower incidence of violence and aggression on the ward via a reduction in the level of arousal and anxiety among inpatients.

DETAILED DESCRIPTION:
Patient aggression and agitation on psychiatric inpatient wards poses a significant problem for both staff and patients, and impairs the therapeutic environment of the ward. Relaxation massage therapy has previously been shown to reduce the level of arousal, stress, anxiety and aggression in adolescents/young adults with various psychiatric disorders including anxiety, depression, conduct disorder and bulimia. This project investigates whether relaxation massage therapy is an effective intervention treatment for the management of arousal and aggression on a young adult inpatient ward.

Two treatment conditions will be assessed at different times on the ward; a) standard (control) treatment as per usual and b) relaxation massage therapy intervention treatment in addition to the standard treatment. Each treatment condition will be implemented for a six-week period. Depending on admission rate, we estimate there will be approximately 50 participants in each treatment group. The massage therapy intervention treatment will consist of daily 20-minute, fully clothed, seated relaxation massage sessions, offered to all consenting patients during their period of hospitalization. We aim to determine whether relaxation massage therapy significantly reduces: i) the level of arousal, stress, anxiety, hostility and aggression in psychiatric inpatients; ii) the frequency and/or severity of aggressive incidents on the ward; iii) the need for sedating medication; iv) the need for patient seclusion and/or restraint; v) the mean duration of hospitalization and vi) the amount of sick leave taken by staff and the associated costs of running the ward. This will be assessed by pre- and post-massage therapy measures of heart rate and salivary cortisol levels; and staff and patient ratings of anxiety, hostility and aggression. The nature, frequency and severity of aggressive incidents on the ward, as well as the use of coercive measures during each treatment condition, will be assessed using the "Staff Observation Aggression Scale-Revised" (SOAS-R). Staff and patient perception of the atmosphere of the ward during each treatment condition will also be assessed using the "Ward Atmosphere Scale".

It is hypothesized that relaxation massage therapy will lead to a lower incidence of violence and aggression on the ward via a reduction in the level of arousal, stress and/or anxiety among inpatients. It is further hypothesized that this will reduce the level of risk for both staff and patients and improve the therapeutic atmosphere of the ward. We also hypothesise that a reduction in aggressive incidents on the ward will be associated with a shorter mean duration of hospitalisation.

ELIGIBILITY:
Inclusion Criteria:

* Admission to the ORYGEN Inpatient Unit

Exclusion Criteria:

* Highly agitated and aggressive patients remaining in a severely aggressive state for more than 24 hours after admission

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 47 (Actual)
Dates: Start 2006-05; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Aggression | 6 weeks
Irritability | 6 weeks
Anxiety | 6 weeks
Depression | 6 weeks
Cortisol levels | 6 weeks

SECONDARY OUTCOMES:
Psychosocial climate | 6 weeks
PRN medication | 6 weeks
Incidence of seclusion or restraint | 6 weeks
Duration of hospitalisation | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Belinda Garner, PhD, Principal Investigator — ORYGEN Research Centre, Department of Psychiatry, University of Melbourne; Lisa Phillips, M.Psych, PhD, Principal Investigator — Department of Psychology, University of Melbourne; Patrick D McGorry, PhD, FRANZP, Study Director — ORYGEN Research Centre , ORYGEN Youth Health, Department of Psychiatry, University of Melbourne
Locations (1):
- ORYGEN Youth Health, Melbourne, Victoria, Australia